CLINICAL TRIAL: NCT01415804
Title: A Randomized Comparison of Strategies for Type B Aortic Dissection - the INvestigation of STEnt-grafts in Aortic Dissection (INSTEAD) Trial
Brief Title: Investigation of Stent-grafts in Aortic Dissection (INSTEAD)
Acronym: INSTEAD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Rostock (Other)
Responsible Party: Christoph A.Nienaber, MD, University of Rostock, Medical School; Dept. of Medicine/Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT00525356; INSTEAD 5 years outcomes (Other Grant/Funding Number: University Hospital Rostock)
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-03

CONDITIONS: Aortic Dissection
Keywords: Dissection; Aorta; Surgery
MeSH Terms: conditions — Aortic Dissection | interventions — Prostheses and Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stentgraft (Active Comparator): Stentgraft
  Interventions: Device: endoprosthesis
- Medical management (No Intervention): Antihypertensive medication
  Interventions: Device: endoprosthesis

INTERVENTIONS:
Device: endoprosthesis — Thoracic aortic stentgraft
  Other Names: Talent endoprosthesis

SUMMARY:
The objective of INSTEAD is to compare long-term (5 years) outcomes of endograft prosthesis versus medical management in patients with dissection of the thoracic aorta.

DETAILED DESCRIPTION:
Patients > 18 years with type B aortic dissection were randomized to either thoracic aortic endoprosthesis (stent-grafting) or antihypertensive management (medical treatment). Only stable patients without spontaneous false lumen thrombosis 14 days after index dissection were considered eligible for study inclusion. Long-term outcome measures included all-cause mortality, aorta-specific mortality and a cluster endpoint (reflecting progression of disease, conversion and additional interventions); the analysis is based on 140 randomized cases followed for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* No contraindication the general anesthesia and ventilation
* Type B aortic dissection that occurred 2-52 weeks prior to randomization
* Diameter of the targeted aortic segment < 6 cm
* Subject or legal guardian understand the nature of teh study and agrees to its provisions on a written informed consent form
* Availability for appropriate follow-up visits during the F/U period of 5 years
* Capability to follow all study requirements

Exclusion Criteria:

* Pregnancy
* Thrombocytopenia
* Ongoing anticoagulation therapy
* Renal failure and/or creatinine > 2,4 mg%
* Complete thrombosis of false lumen
* Cancer likely to cause death within 1 year
* Enrollment in another clinical study
* Unwillingness to cooperate with study procedures or F/U visits

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2002-02; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 5 years post randomization

SECONDARY OUTCOMES:
Aorta-specific mortality | 5 years post randomization
Progression of disease | 5 years
Aortic remodeling | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Nienaber, MD, Principal Investigator — University of Rostock
Locations (1):
- University Hospital Rostock; Heart Center, Rostock, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Background] Nienaber CA, Zannetti S, Barbieri B, Kische S, Schareck W, Rehders TC; INSTEAD study collaborators. INvestigation of STEnt grafts in patients with type B Aortic Dissection: design of the INSTEAD trial--a prospective, multicenter, European randomized trial. Am Heart J. 2005 Apr;149(4):592-9. doi: 10.1016/j.ahj.2004.05.060. PMID 15990739
- [Result] Nienaber CA, Rousseau H, Eggebrecht H, Kische S, Fattori R, Rehders TC, Kundt G, Scheinert D, Czerny M, Kleinfeldt T, Zipfel B, Labrousse L, Ince H; INSTEAD Trial. Randomized comparison of strategies for type B aortic dissection: the INvestigation of STEnt Grafts in Aortic Dissection (INSTEAD) trial. Circulation. 2009 Dec 22;120(25):2519-28. doi: 10.1161/CIRCULATIONAHA.109.886408. Epub 2009 Dec 7. PMID 19996018
- [Derived] Nienaber CA, Kische S, Rousseau H, Eggebrecht H, Rehders TC, Kundt G, Glass A, Scheinert D, Czerny M, Kleinfeldt T, Zipfel B, Labrousse L, Fattori R, Ince H; INSTEAD-XL trial. Endovascular repair of type B aortic dissection: long-term results of the randomized investigation of stent grafts in aortic dissection trial. Circ Cardiovasc Interv. 2013 Aug;6(4):407-16. doi: 10.1161/CIRCINTERVENTIONS.113.000463. Epub 2013 Aug 6. PMID 23922146